CLINICAL TRIAL: NCT06155162
Title: Efficacy of Parent-delivered HuggyPuppy Intervention for Reducing War-related Distress in Young Children
Brief Title: The HuggyPuppy Intervention for War-related Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Michal Kahn, Senior lecturer, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0007481
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Stress Related Disorder
Keywords: psychological intervention; war-related stress; pediatric

STUDY DESIGN:
Who Masked: Participant
Masking Description: Parents will not be masked to the purpose of the intervention, but will be unaware that there are different types of dolls that are being tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Original HuggyPuppy doll (Experimental): The original puppy doll used in Sadeh et al., 2006 is a sad dog with Velcro on its paws will be provided to children allocated to this treatment arm.
  Interventions: Behavioral: The HuggyPuppy Intervention: Original doll
- Monkey with velcro on paws, neutral expression (Experimental): A monkey doll with a neutral expression and with Velcro on its paws will be provided to children allocated to this treatment arm.
  Interventions: Behavioral: The HuggyPuppy Intervention: Monkey doll
- Dog without velcro on paws, neutral expression (Experimental): A puppy doll with a neutral expression and without Velcro on its paws will be provided to children allocated to this treatment arm.
  Interventions: Behavioral: The HuggyPuppy Intervention: Dog without velcro doll
- Bear, smiling (Experimental): A smiling bear doll with a neutral expression and without Velcro on its paws will be provided to children allocated to this treatment arm.
  Interventions: Behavioral: The HuggyPuppy Intervention: Bear doll
- Rabbit, neutral expression (Experimental): A bunny-rabbit doll with a neutral expression and without Velcro on its paws will be provided to children allocated to this treatment arm.
  Interventions: Behavioral: The HuggyPuppy Intervention: Rabbit doll

INTERVENTIONS:
Behavioral: The HuggyPuppy Intervention: Original doll — The HuggyPuppy Intervention, originally designed to alleviate war-related stress in children (Sadeh et al., 2006), is a concise psychosocial intervention featuring a soft plush toy, originally a puppy, accompanied by a 'cover story.' This narrative informs the child that 'Huggy' is seeking care, prompting the child to adopt and comfort the toy. In the parent-delivered version tested in this trial, parents will receive three instructional videos (each lasting 1.5-5 minutes), guiding them on introducing the doll to their child. These videos encourage parents to foster a strong bond between the child and the doll, emphasizing activities such as hugging and expressing emotions through this comforting companion.
  Arms: Original HuggyPuppy doll
Behavioral: The HuggyPuppy Intervention: Monkey doll — The HuggyPuppy Intervention, originally designed to alleviate war-related stress in children (Sadeh et al., 2006), is a concise psychosocial intervention featuring a soft plush toy, originally a puppy, accompanied by a 'cover story.' This narrative informs the child that 'Huggy' is seeking care, prompting the child to adopt and comfort the toy. In this version children receive a plush monkey doll. In the parent-delivered version tested in this trial, parents will receive three instructional videos (each lasting 1.5-5 minutes), guiding them on introducing the doll to their child. These videos encourage parents to foster a strong bond between the child and the doll, emphasizing activities such as hugging and expressing emotions through this comforting companion.
  Arms: Monkey with velcro on paws, neutral expression
Behavioral: The HuggyPuppy Intervention: Dog without velcro doll — The HuggyPuppy Intervention, originally designed to alleviate war-related stress in children (Sadeh et al., 2006), is a concise psychosocial intervention featuring a soft plush toy, originally a puppy, accompanied by a 'cover story.' This narrative informs the child that 'Huggy' is seeking care, prompting the child to adopt and comfort the toy. In this version children receive a plush dog doll, without velcro in palms. In the parent-delivered version tested in this trial, parents will receive three instructional videos (each lasting 1.5-5 minutes), guiding them on introducing the doll to their child. These videos encourage parents to foster a strong bond between the child and the doll, emphasizing activities such as hugging and expressing emotions through this comforting companion.
  Arms: Dog without velcro on paws, neutral expression
Behavioral: The HuggyPuppy Intervention: Bear doll — The HuggyPuppy Intervention, originally designed to alleviate war-related stress in children (Sadeh et al., 2006), is a concise psychosocial intervention featuring a soft plush toy, originally a puppy, accompanied by a 'cover story.' This narrative informs the child that 'Huggy' is seeking care, prompting the child to adopt and comfort the toy. In this version children receive a plush smiling bear doll. In the parent-delivered version tested in this trial, parents will receive three instructional videos (each lasting 1.5-5 minutes), guiding them on introducing the doll to their child. These videos encourage parents to foster a strong bond between the child and the doll, emphasizing activities such as hugging and expressing emotions through this comforting companion.
  Arms: Bear, smiling
Behavioral: The HuggyPuppy Intervention: Rabbit doll — The HuggyPuppy Intervention, originally designed to alleviate war-related stress in children (Sadeh et al., 2006), is a concise psychosocial intervention featuring a soft plush toy, originally a puppy, accompanied by a 'cover story.' This narrative informs the child that 'Huggy' is seeking care, prompting the child to adopt and comfort the toy. In this version children receive a plush rabbit doll, with a neutral expression. In the parent-delivered version tested in this trial, parents will receive three instructional videos (each lasting 1.5-5 minutes), guiding them on introducing the doll to their child. These videos encourage parents to foster a strong bond between the child and the doll, emphasizing activities such as hugging and expressing emotions through this comforting companion.
  Arms: Rabbit, neutral expression

SUMMARY:
This clinical trial will test the efficacy of parent-delivered HuggyPuppy Intervention in alleviating war-related stress in children aged 3-8 during the Gaza-Israel war. Moreover, it will test whether the type of doll provided moderates the efficacy of the intervention. Children will be provided a doll ('Huggy') of to their homes or places of shelter, and asked to take care of it. Five different types of dolls will be randomly assigned to children. Pre-intervention, parents will complete a brief questionnaire asking about the child's past week stress symptoms, and exposure to traumatic war-experiences. Three weeks following the intervention, parents will be asked to complete a post-intervention questionnaire, asking about the child's symptoms, their own anxiety, depression, and stress, as well as their use of the intervention.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test the efficacy of parent-delivered HuggyPuppy Intervention in alleviating war-related stress in children aged 3-8 during the Gaza-Israel war. The trial also aims to examine whether the type of doll provided moderates the efficacy of the intervention, and whether parent and child attachment to the doll and adherence to the intervention are associated with its outcomes.

Participants will be 160 children aged 3-8 from across Israel, whose parents perceive them to be distressed due to the war. Parents will undergo a brief phone interview to confirm the child's age and distress level. Subsequently, parents will be directed to complete a concise online survey, detailing their child's stress symptoms over the past week and exposure to traumatic war experiences. Demographic information, such as parent marital status, will also be collected.

The HuggyPuppy Intervention will then be delivered to all children via their parents. This brief psychosocial intervention was originally developed to reduce war-related stress in children (Sadeh et al., 2006). It involves a soft plush toy - originally a puppy - provided to the child along with a 'cover story', telling the child that 'Huggy' (the puppy) is far from home and looking for someone to look after it. The child is then asked to adopt Huggy, and take care of it when it is sad and lonely.

Children will be randomly assigned to receive one of five different types of dolls (dog with Velcro in palms, dog without Velcro in palms, monkey with Velcro in palms, bear, and rabbit). The doll will be delivered to their homes or places of shelter. During the course of 1 week of intervention, parents will receive three instructional videos (each lasting 1.5-5 minutes), guiding them on how to introduce the doll to their child. They will be encouraged to nurture a bond between the child and the doll, promoting activities like hugging and expressing emotions through it. Three weeks after the intervention, parents will be requested to complete a post-intervention questionnaire. This questionnaire will cover the child's symptoms, as well as the parent's anxiety, depression, and stress levels. Additionally, parents will provide feedback on their adherence to and experiences with the intervention.

The expected results of this study will provide empirical evidence on the effectiveness of the parent-delivered HuggyPuppy Intervention in ameliorating war-related stress in young children. Moreover, the study aims to enhance our understanding of potential moderating factors, such as the type of doll provided, and shed light on the crucial role of parent and child attachment to the intervention, offering valuable insights for the development of targeted interventions in the context of conflict-related stress.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 3-8 years old
* Parents perceive child to be in distress due to the war (<1 on a scale from 1-5, 1=not at all distressed, and 5=very high distress).
* Parent proficiency in Hebrew

Exclusion Criteria:

* N/A

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Stress reactions | This measure will be completed by parents at pre- and 3-weeks post-intervention.
  A stress reaction checklist (SRCL) will be used to assess children's level of stress-related symptoms. These include 15 items, such as "excessive crying", "experiencing nighttime awakenings or nightmares", and "frequently speaks about death". A general item pertaining to the child's level of distress on a 5-point scale will also be administered.

SECONDARY OUTCOMES:
Intervention adherence and satisfaction | Post-treatment only
  Parents will complete a series of questions about their use and experience of the intervention. Items will refer to child attachment to the doll, and parent perception of and compliance with instructions (e.g., watching all 3 instructional videos), as well as their satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, analysis plan, all forms and measures, and the clinical report will be available to any requesting party, that plans to use this for educational or research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available upon completion of recruitment.
Access Criteria: Request from Primary Investigator